CLINICAL TRIAL: NCT06251011
Title: Effects of Physiotherapy Via Telerehabilitation on Cardiopulmonary, Physical, and Psychological Functions in Patients With COVID-19: A Randomized Controlled Trial
Brief Title: Effects of Physiotherapy Via Telerehabilitation in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulabhorn Hospital (Other)
Responsible Party: Principal Investigator, Pooriput Waongenngarm, PT, PhD, Assistant Professor, Chulabhorn Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC014/2565
Record Dates: First submitted 2024-02-07; First posted 2024-02-09 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: COVID-19; Long COVID-19; Cardiopulmonary Function; Physical Function
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Receive an advice and a leaflet for cardiopulmonary rehabilitation.
- Physiotherapy group (Experimental): Receive the physical therapy training via video call (Pulmonary training, Calisthenic exercise, Upper and lower limbs strengthening exercise, Core stabilizer exercise, Aerobic exercise) at day 3, 6, 9, 12, 16, and 21 after positive in COVID-19 testing and also receive advise and a leaflet for cardiopulmonary rehabilitation.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — 1. Physical therapy training via video call
  2. An advise and a leaflet for cardiopulmonary rehabilitation
  Arms: Physiotherapy group

SUMMARY:
This study aims to evaluate the effects of Physiotherapy Via Video Calls on Cardiopulmonary Functions, Physical Function, Cognitive Function, Activity Daily Livings, and Quality of Life in Patients With COVID-19.

DETAILED DESCRIPTION:
A 2-armed, parallel-group, randomized controlled trial was conducted at Chulabhorn Hospital, Thailand on a convenience sample of patients who tested positive for COVID-19 using RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-60 years old
* Positive in COVID-19 testing
* Good communication and understanding
* Independent mobility

Exclusion Criteria:

* Cannot complete the study protocol

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary function | at day 28 and 90 after positive in COVID-19 testing
  using Cardiopulmonary exercise testing (CPET)
Patient's quality of life | at day 3 and 21 after positive in COVID-19 testing
  using the The World Health Organization Quality of Life (WHOQOL-BREF-THAI) 26 items; the final score ranges from 24-120; higher score means participants satisfied with the quality of life.
Functional capacity | at day 3 and 21 after positive in COVID-19 testing
  using Duke Activity status index The final score ranges between zero and 58.2 points; The higher the score, the better the functional capacity.
Anxiety and depression | at day 3 and 21 after positive in COVID-19 testing
  using Hospital Anxiety and Depression Scale (HADS) The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Insomnia | at day 3 and 21 after positive in COVID-19 testing
  using Insomnia Severity Index (ISI) The final score ranges between zero and 28 points. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Cognitive function | at day 3 and 21 after positive in COVID-19 testing
  using Thai Mental State Examination The final score ranges between zero and 30 points. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
Muscle strength | at day 3 and 21 after positive in COVID-19 testing
  using 1-minute sit to stand

CONTACTS AND LOCATIONS:
Overall Officials: Pooriput Waongenngarm, PhD, Principal Investigator — Chulabhorn Royal Academy
Locations (1):
- Chulabhorn hospital, Lak Si, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Due to the ethical restriction, investigators cannot share any individual participant data.